CLINICAL TRIAL: NCT07084311
Title: An Open-label, Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for ATN1 Mutation Associated Dentatorubral-pallidoluysian Atrophy (DRPLA)
Brief Title: Personalized Antisense Oligonucleotide for A Single Participant With ATN1 Gene Mutation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Hawaii Pacific Neuroscience (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081366
Record Dates: First submitted 2025-05-08; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Dentatorubral-Pallidoluysian Atrophy
MeSH Terms: conditions — Myoclonic Epilepsies, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-ATN1-002

INTERVENTIONS:
Drug: nL-ATN1-002 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with dentatorubral-pallidoluysian atrophy (DRPLA) due to a heterozygous pathogenic CAG trinucleotide expansion in ATN1

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with DRPLA due to a heterozygous pathogenic CAG trinucleotide expansion in ATN1

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Clinical phenotype and neuroimaging consistent with a diagnosis of ATN1 mutation associated Dentatorubral-pallidoluysian atrophy (DRPLA).
* Documented genetic mutation in ATN1.

Exclusion Criteria:

* Participant has any known contraindication to or unwillingness to undergo lumbar puncture.
* Use of investigational medication within 5 half-lives of the drug at enrollment.
* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.

Ages: 29 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Seizures | Baseline to 24 months
  Change in seizure length from baseline to every 3 months post nL-ATN1-002 administration as measured by routine electroencephalography (EEG)
Seizures | Baseline to 24 months
  Change in seizure frequency and seizure medication use from baseline to every 3 months post nL-ATN1-002 administration as measured by seizure tracking (reported with seizure dates and use of seizure medication).

SECONDARY OUTCOMES:
Quality of Life and Caregiver Burden | 24 months
  Change in quality of life and caregiver burden from baseline to 6-, 12-, 18-, and 24- months post nL-ATN1-002 administration as measured by the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD)
Health Status | 24 months
  Change in health issues from baseline to 6-, 12-, 18-, and 24-months post nL-ARN1-002 administration as measured by the Caregiver Priorities - Comorbidities and Health Evaluation Checklist (CPCHECKlist)
Incidence and Severity of Treatment Emergent Adverse Events [Safety and Tolerability] | 24 months
Incidence of Treatment-Emergent Abnormalities in Physical and Neurological Exams [Safety and Tolerability] | 24 months
Incidence of Treatment-Emergent Abnormalities in Safety Labs (CSF, chemistry, hematology, coagulation, and urinalysis) [Safety and Tolerability] | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hawaii Pacific Neuroscience, Honolulu, Hawaii, United States